CLINICAL TRIAL: NCT00823069
Title: A Randomized, Double-Blind Study Comparing Safety and Tolerability of Perlane® With and Without Addition of 0.3% Lidocaine HCL During Correction of Nasolabial Folds
Brief Title: Safety Study That Compares Perlane to Perlane With Lidocaine (Perlane-L) While Correcting Wrinkles in the Area Around Your Nose
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medicis Global Service Corporation (Industry)
Collaborators: Q-Med Scandinavia, Inc. (Industry)
Responsible Party: Mary Sanstead, Clinical Study Manager, Medicis Global Services
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MA-1400-03
Record Dates: First submitted 2009-01-14; First posted 2009-01-15 (Estimated); Results first posted 2010-11-30 (Estimated); Last update posted 2010-11-30 (Estimated); Status verified 2010-11

CONDITIONS: Nasolabial Folds
Keywords: Correction of Nasolabial Folds

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Perlane and Perlane-L (Other): This is a split-face design injecting both Perlane and Perlane-L injectable gels, administered once. Each subject received Perlane-L on one side of the face, and Perlane on the other. Subjects were blinded to which side of their face receive Perlane or Perlane-L. The study was randomized and treatments successive.
  Interventions: Device: Perlane and Perlane-L

INTERVENTIONS:
Device: Perlane and Perlane-L — This is a split face design and each subject received both Perlane-L and Perlane. Treatments were blinded, randomized, and successive.
  Other Names: Each subject received both Perlane-L and Perlane.

SUMMARY:
Safety study that compares Perlane to Perlane with Lidocaine while correcting wrinkles in the area around your nose.

DETAILED DESCRIPTION:
This is a split-face design. All 60 subjects receive Perlane on one side of their face, and Perlane-L on the other. Subjects and the investigator is blinded to which side of face receives which product. These are one time injections.

ELIGIBILITY:
Inclusion Criteria:

* Same Wrinkle Severity Rating Scale score at both Nasolabial Folds (either both Moderate [3] or both Severe [4])

Exclusion Criteria:

* Active or chronic skin disease, inflammation or related conditions, near or on the Nasolabial Folds
* Subjects who had undergone procedures based on active dermal response (e.g., laser or chemical peeling procedures) within 6 months prior to study entry
* Use of any facial tissue augmenting therapy with non-permanent filler or aesthetic facial surgical therapy within 9 months prior to study entry
* Permanent implant placed in the Nasolabial Fold area

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-01; Primary Completion 2009-03 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Sanstead, Study Chair — Medicis Global Pharmaceutical
Locations (3):
- United States (3):
  - Coral Gables, Florida
  - Hunt Valley, Maryland
  - Mount Cisco, New York

RESULTS

PARTICIPANT FLOW:
Groups:
- Perlane-L and Perlane: Split face design with each subject receiveing Perlane on one side of the face and Perlane-L on the other.
Period: Overall Study
Arm/Group | Perlane-L and Perlane
Started | 60
Completed | 60
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Perlane and Perlane-L: Split face design with each subject receiveing Perlane on one side of the face and Perlane-L on the other.
Arm/Group | Perlane and Perlane-L
Number analyzed (Participants) | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 60
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 53.4 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 60

OUTCOME MEASURES:

1. Primary Outcome: Treatment Difference in VAS (Perlane Side - Perlane-L Side) With Difference in VAS >= 10 mm
Time Frame: After Injection on Day of Treatment
Population: This is a split-face design. Perlane and Perlane with Lidocaine was applied to different sides of the subject's face. A total of 60 subjects received both products. The study evaluated which side of the face has less pain, as measured by the Visual Analogue Scale (VAS). Least pain on VAS scale is at 0 mm mark and worst pain is 100 mm mark.
Measure: Number (95% Confidence Interval); unit: Participants
Arm/Group | Perlane-L and Perlane
Number analyzed (Participants) | 60
Participants | 95 [86.1 to 99]

2. Secondary Outcome: Number of Subjects Showing Wrinkle Improvement at Day 14
Description: This measure was performed by the validated GAIS tool (Global Asthetic Improvement Scale). The GAIS was completed by the participant at day 14. The GAIS is a qualitative 5 point scale evaluating Aesthetic Improvement (0=worse, 1=no change, 2=Improved, 3=Much Improved, 4=very much improved). Treatment success is defined as at least a one grade improvement (2, 3, or 4) from pre-treatment.
Time Frame: 14 days after treatment when compared to baseline
Measure: Number; unit: Participants
Groups:
- Perlane-L; Perlane: Split face design with each subject receiving Perlane on one side of the face and Perlane-L on the other. After treatments the patient scores pain experienced on a 2 VAS scales. One VAS represents pain on the left side of face, and the other VAS for the right side of the face. Least pain on VAS is at the 0 mm mark, and worst pain is at the 100 mm mark. Objective is to calculate the proportion of subjects that had a within-subject difference in the VAS (Perlane minus Perlan-L) of at least 10 mm at injection together with a 95% confidence interval. The objective was to show that the confidence interval lay above 50%.
Arm/Group | Perlane-L | Perlane
Number analyzed (Participants) | 60 | 60
Participants | 57 | 58

ADVERSE EVENTS:
Arm/Group | Perlane-L | Perlane
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/60
Other Adverse Events (participants affected / at risk) | 60/60 | 60/60
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Perlane-L (N=60) | Perlane (N=60)
Bruising (General disorders) | 36 (36) | 33 (33)
Redness (General disorders) | 34 (34) | 31 (31)
Swelling (General disorders) | 42 (42) | 39 (39)
Pain (General disorders) | 28 (28) | 26 (26)
Tenderness (General disorders) | 50 (50) | 49 (49)
Itching (General disorders) | 16 (16) | 12 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days